CLINICAL TRIAL: NCT06398132
Title: Thalidomide-Related Investigation on Understanding and Managing Pain for Thalidomide Survivors
Brief Title: Understanding and Managing Pain for Thalidomide Survivors
Acronym: TRIUMPH-TS
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: The Thalidomide Trust (Unknown)
Responsible Party: Principal Investigator, Vasileios Georgopoulos, Principal Investigator, University of Nottingham
Other Study IDs: 112-0224
Record Dates: First submitted 2024-04-24; First posted 2024-05-03 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Pain, Chronic; Pain
Keywords: Thalidomide; Pain; Pain Management; Intervention Development
MeSH Terms: conditions — Chronic Pain; Pain; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Thalidomide Survivors: The group will include Thalidomide Survivors (n=120), who are beneficiaries of the Thalidomide Trust and receive Usual Care for the management of their pain. Usual Care includes among others, over-the-counter or prescribed painkillers, treatment modalities such as physiotherapy and/or psychotherapy, privately accessed or via the National Health Service, exercise, etc.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Usual Care — Usual Care includes among others, over-the-counter or prescribed painkillers, treatment modalities such as physiotherapy and/or psychotherapy, privately accessed or via the National Health Service, exercise, etc.

SUMMARY:
Aim: To explore the pain experience of Thalidomide survivors and propose an effective pain management service, tailored to meet the unique needs of this population.

Background: Approximately 400 thalidomide survivors live in the UK, who are also beneficiaries of the Thalidomide Trust. Such individuals have been mainly born with upper or lower limb problems, but some also experience sight, hearing, or speaking difficulties. Most tend to experience additional problems, acquired after birth, including persistent muscle or joint pain as well as mental health problems. Such conditions may reduce the quality of life of thalidomide survivors, who face significant difficulties in accessing healthcare services or receiving effective treatment. Specialist services such as pain management are not easily available to thalidomide survivors. Providers' lack of understanding or flexibility to treat populations with unique needs, and geographical or financial barriers have been considered as possible reasons.

Methods: This is a cross-sectional observational study. Thalidomide survivors, who are also beneficiaries of the Thalidomide Trust, will be offered a questionnaire booklet to fill, featuring questionnaires aiming to explore their pain experience (0-10 Pain Numerical Rating Scale, Central Aspects of Pain, painDETECT, Widespread Pain Index), mental health (Hospital Anxiety and Depression Scale), beliefs (Pain Catastrophizing, Tampa Scale of Kinesiophobia), quality of life (EQ-5D-5L), disability (Health Assessment Questionnaire), sleep (Athens Insomnia Scale), and medicines use (Pain Medication Attitude Questionnaire). Linear regression modelling will explore the factors that best explain the overall pain experience of Thalidomide Survivors.

Impact: The research will inform how thalidomide survivors might gain access to an evidence-based pain management service designed specifically for them, which will improve their quality of life.

DETAILED DESCRIPTION:
Between 1958 and 1961, Thalidomide was widely prescribed in the UK as a safe, non-addictive sedative and tranquiliser. Despite being marketed as an entirely safe treatment for the discomforts of pregnancy (including morning sickness), Thalidomide caused serious damage to the unborn child when taken during the first trimester. Foetal damage typically included upper and/or lower limb malformation (total limb absence, missing bones, etc), eye, ear and facial damage (damaged ears, narrow ear canals, small or damaged eyes, restricted eye movement and facial palsy), and malformation of internal organs (heart, urinary and alimentary tracts, and reproductive organs). Collectively, such birth defects are referred to as Thalidomide Embryopathy or Thalidomide Syndrome. A charitable trust - the Thalidomide Children's Trust (now the Thalidomide Trust), was established to oversee compensation payments from Distillers to those children affected by Thalidomide in the UK.

Thalidomide survivors experience significantly worse physical and mental health than the general population of the same age, demonstrating a wide range of secondary health problems, in particular chronic musculoskeletal pain, which is the most reported symptom, as well as movement restrictions, and mental disorders. Such health problems impair the ability of these individuals to remain fully independent, and negatively impact on their health-related quality of life as they limit their overall ability to adopt an active lifestyle and engage or access potentially beneficial treatments.

Thalidomide survivors form a unique, underrepresented, and disadvantaged group of people who must overcome a number of additional barriers in order to receive appropriate care. Compared with non-Thalidomide age-matched populations, Thalidomide survivors demonstrate higher prevalence of pain and disability. However, most comparisons have been done with members of the general population. Thalidomide Trust beneficiaries with lived experience of chronic pain might share features with other populations with chronic musculoskeletal pain (e.g., Fibromyalgia, Rheumatoid Arthritis, Chronic Low Back Pain), such as reluctance to take tablets due to their formative experience with medicines, poor experiences from exposure to multiple interventions and surgeries, and difficult experiences with health care professionals who seem not to understand or often dismiss their unique and complex needs. Despite the prevalence of shared features, Thalidomide survivors might also experience unique issues that are not shared with other populations with chronic pain. Whilst effective pain management has become more accessible to some populations with chronic musculoskeletal pain, for Thalidomide survivors, inequity persists. Novel research, investigating the lived experience of pain by Thalidomide survivors, is needed explore potential barriers in pain management of Thalidomide Survivors.

To address this gap in literature the project aims to define the pain experience of beneficiaries. This cross-sectional observational study entails a questionnaire booklet designed to collect numerical and categorical data about the experience of pain by Thalidomide survivors as well as the impact of pain on their lives and overall wellbeing. To ensure that participants adequately represent Thalidomide survivors as a unique population, a purposive sampling strategy will be followed.

Distinct categories of pain have been identified in the general population, such as neuropathic pain, nociplastic pain, or chronic primary pain. The project will quantitatively, via collection of new primary data, explore whether these categories can be also identified in Thalidomide survivors, whether one or more category is more common than others, and whether there is a unique 'Thalidomide pain' category. A combination of different sets of criteria developed by the International Association for the Study of Pain (IASP) and patient reported outcome measures, namely Central Aspects of Pain (CAP) and painDETECT, will be used for categorising.

All beneficiaries of the Thalidomide Trust can potentially be recruited (n≈400). However, past pain-related research exploring combinations of biopsychosocial variables and pain intensity 2 has shown that with estimated variation of 40% (R2=0.40) and an estimated number of independent variables (5 to 7) to be included in regression analyses, 120 individuals are considered sufficient to power the study and explain 38-49% of the variance in the regression model. Calculations are based on the estimated squared multiple correlation-coefficient (R2) [10].

Regression analyses will explore whether certain factors, potentially identified also as barriers in the qualitative aspect of the WP, are associated with the experience of pain.

ELIGIBILITY:
Inclusion Criteria:

* Be beneficiaries of the Thalidomide Trust
* Be able to communicate in English or via using the British Sign Language as all interview questions and questionnaires are designed in the English language

Exclusion Criteria:

* Inability to give informed consent due to cognitive impairment or otherwise - (capacity levels are already established under General Practitioner (GP) care)
* Inability to understand key aspects of the study due to cognitive impairment or otherwise
* Giving history of critical or terminal co-morbidities such as cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Thalidomide survivors experience significantly worse physical and mental health than the general population of the same age, demonstrating a wide range of secondary health problems, in particular chronic musculoskeletal pain, which is the most reported symptom, as well as movement restrictions, and mental disorders. Such health problems impair the ability of these individuals to remain fully independent, and negatively impact on their health-related quality of life as they limit their overall ability to adopt an active lifestyle and engage or access potentially beneficial treatments. Thalidomide survivors form a unique, under-represented, and disadvantaged group of people who must overcome a number of additional barriers in order to receive appropriate care.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Central Aspects of Pain (CAP) [Modified] | Through study completion, an average of 1 year
  A tool featuring 7 questions and a body manikin, designed to indicate distinct central pain mechanisms. Higher scores indicate dominance of central mechanisms in the overall pain experience. A modified version without the manikin [the tick-box choices for each body site used in CAP will be applied] will be used out of respect to Thalidomide Survivors. A modified version replacing the manikin with tick-box available for each body site will be used out of respect to Thalidomide Survivors.
painDETECT (PDQ) [Modified] | Through study completion, an average of 1 year
  A tool featuring 9 questions and a body manikin, designed to indicate neuropathic mechanisms for pain. Higher scores indicate dominance of neuropathic mechanisms in the overall pain experience. A modified version without the manikin [the tick-box choices for each body site used in CAP will be applied] will be used out of respect to Thalidomide Survivors.
Widespread Pain Index (WPI) [Modified] | Through study completion, an average of 1 year
  A tool featuring a body manikin, 3 symptom severity scales, measuring fatigue, waking up unrefreshed, and cognitive dysfunction, and a somatic symptoms list. Higher scores indicate dominance of central mechanisms and increased likelihood of a positive diagnosis of fibromyalgia. A modified version without the manikin [the tick-box choices for each body site used in CAP will be applied] will be used out of respect to Thalidomide Survivors.

SECONDARY OUTCOMES:
0-10 Numerical Rating Scale (NRS) | Through study completion, an average of 1 year
  Three simple 0-10 numerical rating scales (min: 0 = no pain, max: 10 = extreme pain) asking to rate pain severity now, strongest pain over the last week, and average pain over the last week.Higher scores mean higher pain severity.
Hospital Anxiety and Depression Scale (HADS) | Through study completion, an average of 1 year
  HADS is comprised by 7 questions about depression (min: 0, max: 21) and 7 questions about anxiety (min: 0, max: 21). Each component yields a distinct score. Higher scores indicate higher levels of symptoms of depression and anxiety.
Pain Catastrophizing Scale (PCS) | Through study completion, an average of 1 year
  PCS is comprised by 13 questions aiming to capture thoughts people have about their pain (min: 0, max: 52). Higher score indicates higher levels of catastrophizing.
Tampa Scale of Kinesiophobia (TSK) | Through study completion, an average of 1 year
  TSK is comprised by 17 questions aiming to thoughts and fears they have developed about their pain, as well as movements associated with it (min: 17, max: 68). Higher score indicates higher levels of kinesiophobia
EuroQoL 5-Dimensions 5-Levels (EQ-5D-5L) | Through study completion, an average of 1 year
  EQ-5D-5L is comprised by 5 dimensions (Mobility, Self-care, Usual Activities, Pain/Discomfort, Anxiety/Depression), each comprised by 5 distinct levels of severity. An index score (min: 0.0, max: 1.0) is produced that indicates quality of life for each individual. Additionally, a 0-100 Visual Analogue Scale (min: 0, max: 100) provides insight about overall health. Higher scores indicate better overall health.
Health Assessment Questionnaire - Disability (HAQ-DI) | Through study completion, an average of 1 year
  HAQ-DI is comprised by distinct dimensions (Dressing & Grooming, Arising, Eating, Walking, Aids or Devices, Hygiene, Reach, Grip, Activities, and Help from Another Person) (min:0, max: 3 on each category). The eight category scores are averaged into an overall HAQ-DI score on a scale from 0 (no disability) to 3 (completely disabled). Higher score indicates higher levels of disability.
Athens Insomnia Scale (AIS) | Through study completion, an average of 1 year
  AIS is comprised by 8 questions (min: 0, max: 28) about sleeping habits and sleep quality. Higher score indicates higher levels of sleep disturbance and insomnia.
Pain Medication Attitude Questionnaire (PMAQ) | Through study completion, an average of 1 year
  PMAQ is comprised by 7 domains [Addiction (min: 0, max: 25), Need (min: 0, max: 40), Scrutiny (min: 0, max: 40), Side effects (min: 0, max: 35), Tolerance (min: 0, max: 30), Mistrust of Doctors (min: 0, max: 35), Withdrawal (min: 0, max: 30) reflected in 47 questions about medicines use and attitudes towards them. Higher score within each domain indicates higher levels of sub-optimal medicines use and negative attitudes towards them.

CONTACTS AND LOCATIONS:
Overall Officials: Vasileios Georgopoulos, PhD, Principal Investigator — University of Nottingham; David A. Walsh, PhD, Study Chair — University of Nottingham; Daniel F. McWilliams, PhD, Study Chair — University of Nottingham; Fionna Moffatt, PhD, Study Chair — University of Nottingham; Holly Blake, PhD, Study Chair — University of Nottingham
Locations (1):
- Clinical Sciences Building - City Hospital Campus, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Agreement is already in place for anonymised raw data of all study outcomes to be shared with the Thalidomide Trust. Agreement is already in place for anonymised raw dat of the painDETECT questionnaire to be shared with IQVIA, who is the provider of the tool.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For the Thalidomide Trust, after analysis is completed. For IQVIA, as soon as recruitment ends and data input is complete.
Access Criteria: A separate data sharing agreement will need to be signed, as per the policies of the University of Nottingham, with each party wishing to access the data of this study.
URL: https://www.nottingham.ac.uk/library/documents/research/data-management-plan-resources/data-sharing-guidance/2022datasharingguidance.pdf

REFERENCES:
- [Background] Smithells RW, Newman CG. Recognition of thalidomide defects. J Med Genet. 1992 Oct;29(10):716-23. doi: 10.1136/jmg.29.10.716. No abstract available. PMID 1433232
- [Background] Niecke A, Peters KM, Alayli A, Lungen M, Pfaff H, Albus C, Samel C. Health-related quality of life after 50 years in individuals with thalidomide embryopathy: Evidence from a German cross-sectional survey. Birth Defects Res. 2022 Aug 1;114(13):714-724. doi: 10.1002/bdr2.2051. Epub 2022 Jun 4. PMID 35666030
- [Background] Ghassemi Jahani SA, Karlsson J, Brisby H, Danielsson AJ. Health-related quality of life and function in middle-aged individuals with thalidomide embryopathy. J Child Orthop. 2016 Dec;10(6):691-703. doi: 10.1007/s11832-016-0797-6. Epub 2016 Nov 16. PMID 27854003
- [Background] Jankelowitz SK, Spies JM, Burke D. Late-onset neurological symptoms in thalidomide-exposed subjects: a study of an Australasian cohort. Eur J Neurol. 2013 Mar;20(3):509-514. doi: 10.1111/ene.12005. Epub 2012 Oct 18. PMID 23078293
- [Background] Vargesson N, Hooper G, Giddins G, Hunter A, Stirling P, Lam W. Thalidomide upper limb embryopathy - pathogenesis, past and present management and future considerations. J Hand Surg Eur Vol. 2023 Sep;48(8):699-709. doi: 10.1177/17531934231177425. Epub 2023 May 24. PMID 37226469
- [Background] Newbronner E, Glendinning C, Atkin K, Wadman R. The health and quality of life of Thalidomide survivors as they age - Evidence from a UK survey. PLoS One. 2019 Jan 16;14(1):e0210222. doi: 10.1371/journal.pone.0210222. eCollection 2019. PMID 30650111
- [Background] Nijs J, George SZ, Clauw DJ, Fernandez-de-Las-Penas C, Kosek E, Ickmans K, Fernandez-Carnero J, Polli A, Kapreli E, Huysmans E, Cuesta-Vargas AI, Mani R, Lundberg M, Leysen L, Rice D, Sterling M, Curatolo M. Central sensitisation in chronic pain conditions: latest discoveries and their potential for precision medicine. Lancet Rheumatol. 2021 May;3(5):e383-e392. doi: 10.1016/S2665-9913(21)00032-1. Epub 2021 Mar 30. PMID 38279393
- [Background] Nijs J, Lahousse A, Kapreli E, Bilika P, Saracoglu I, Malfliet A, Coppieters I, De Baets L, Leysen L, Roose E, Clark J, Voogt L, Huysmans E. Nociplastic Pain Criteria or Recognition of Central Sensitization? Pain Phenotyping in the Past, Present and Future. J Clin Med. 2021 Jul 21;10(15):3203. doi: 10.3390/jcm10153203. PMID 34361986
- [Background] Chronic pain (primary and secondary) in over 16s: assessment of all chronic pain and management of chronic primary pain. London: National Institute for Health and Care Excellence (NICE); 2021 Apr 7. Available from http://www.ncbi.nlm.nih.gov/books/NBK569960/ PMID 33939353
- [Background] Knofczynski GT, Mundfrom D. Sample sizes when using multiple linear regression for prediction. Educational and Psychological Measurement. 2008;68(3):431-442.